CLINICAL TRIAL: NCT02437071
Title: Single Arm Phase II Study to Assess the Efficacy of Pembrolizumab Plus Radiotherapy or Ablation in Metastatic Colorectal Cancer Patients
Brief Title: Assess the Efficacy of Pembrolizumab Plus Radiotherapy or Ablation in Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-069
Record Dates: First submitted 2015-04-22; First posted 2015-05-07 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Radiotherapy; Ablation; Pembrolizumab; 15-069; Metastatic Colorectal Cancer Patients
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Radiotherapy; Radiofrequency Ablation

ARMS (2):
- Pembrolizumab Plus Radiotherapy (Experimental): pembrolizumab plus RT in subjects with metastatic CRC who are undergoing RT as standard therapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy
- Pembrolizumab Plus Ablation (Experimental): pembrolizumab plus ablation in subjects with metastatic CRC who are undergoing ablation as standard therapy
  Interventions: Drug: Pembrolizumab; Procedure: Radiofrequency ablation

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered as a 30 minute IV infusion (every effort should be made to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
Radiation: Radiotherapy
  Arms: Pembrolizumab Plus Radiotherapy
Procedure: Radiofrequency ablation
  Arms: Pembrolizumab Plus Ablation

SUMMARY:
The radiation therapy or ablation that the patient received as standard therapy treated only the tumors that were radiated or ablated. Radiation therapy or ablation plus pembrolizumab might lead to a stronger immune response that may control or destroy tumors that did not receive radiation therapy or ablation. The purpose of this study is to find out what effects, good and/or bad, pembrolizumab has on the patient, and the cancer that did not receive radiation therapy or ablation.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Histologically- or cytologically- confirmed CRC.
* Metastatic or recurrent CRC
* Subjects have received two or more standard available therapies known to prolong survival and for which they would be considered eligible. Such therapies should include regimens containing oxaliplatin and irinotecan in combination with a fluoropyrimidine if appropriate (e.g., FOLFOX and FOLFIRI or their variants).
* At least one tumor for which palliative RT is considered appropriate standard therapy (cohort 1); or, at least one tumor for which palliative ablation is considered appropriate standard therapy (cohort 2).
* At least one index lesion that will not undergo RT or ablation, and which is measurable based on RECIST 1.1.
* Be ≥ 18 years of age on day of signing informed consent. Consent for tumor biopsies and blood draws for research purposes.
* Consent for use of available archived tissue for research purposes.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 6.1, all screening labs should be performed within 6 weeks of treatment initiation.

Hematological

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL Renal
* Serum creatinine OR Measured or calculated* creatinine clearance (GFR can also be used in place of creatinine or CrCl)
* ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR
* Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT)
* ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

  * Creatinine clearance should be calculated per institutional standard.
* Female subject of childbearing potential should have a negative serum pregnancy within 2 weeks prior to starting radiation therapy or undergoing ablation.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 9.5.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  ° Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Mendonca Gorgulho C, Krishnamurthy A, Lanzi A, Galon J, Housseau F, Kaneno R, Lotze MT. Gutting it Out: Developing Effective Immunotherapies for Patients With Colorectal Cancer. J Immunother. 2021 Feb-Mar 01;44(2):49-62. doi: 10.1097/CJI.0000000000000357. PMID 33416261
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab Plus Radiotherapy: pembrolizumab plus RT in subjects with metastatic CRC who are undergoing RT as standard therapy
  Pembrolizumab: Pembrolizumab will be administered as a 30 minute IV infusion (every effort should be made to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
  Radiotherapy
- Pembrolizumab Plus Ablation: pembrolizumab plus ablation in subjects with metastatic CRC who are undergoing ablation as standard therapy
  Pembrolizumab: Pembrolizumab will be administered as a 30 minute IV infusion (every effort should be made to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
  Radiofrequency ablation
Period: Overall Study
Arm/Group | Pembrolizumab Plus Radiotherapy | Pembrolizumab Plus Ablation
Started | 25 | 9
Completed | 24 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Plus Radiotherapy | Pembrolizumab Plus Ablation | Total
Number analyzed (Participants) | 25 | 9 | 34
Age, Continuous [Mean (Full Range); unit: years] | 60 [18 to 80] | 59 [35 to 72] | 59.7 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 4 | 16
  Unknown or Not Reported | 13 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 22 | 7 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: If at the end of the study ≥3 tumor responses per RECIST 1.1 are observed in a cohort, then further investigation of pembrolizumab plus RT and/or pembrolizumab plus ablation will be considered worthwhile. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) no PR - no Progressive Disease (PD); Progressive Disease (PD) >=20% increase sum of longest diameters of the target lesions (SLD) compared to smallest SLD in study or progression of non-target lesions or new lesions
Time Frame: approximately 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus Radiotherapy | Pembrolizumab Plus Ablation
Number analyzed (Participants) | 24 | 9
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 1
  Stable Disease | 5 | 1
  Progressive Disease | 18 | 7

2. Secondary Outcome: Number of Participants With Toxicities
Description: All recorded toxicity will be listed and tabulated by system organ class, preferred term and treatment. Any significant vital signs and clinical laboratory test results will be listed and summarized. Any significant physical examination findings, and clinical laboratory results will be listed. Will be recorded according to "Common Terminology Criteria for Adverse Events" V4.0 (CTCAE).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus Radiotherapy | Pembrolizumab Plus Ablation
Number analyzed (Participants) | 24 | 9
Participants | 24 | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pembrolizumab Plus Radiotherapy | Pembrolizumab Plus Ablation
All-Cause Mortality (participants affected / at risk) | 21/25 | 9/9
Serious Adverse Events (participants affected / at risk) | 21/25 | 9/9
Other Adverse Events (participants affected / at risk) | 25/25 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radiotherapy (N=25) | Pembrolizumab Plus Ablation (N=9)
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastric Obstruction (Gastrointestinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Death NOS (General disorders) | 21 | 9
Abdominal Infection (Infections and infestations) | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radiotherapy (N=25) | Pembrolizumab Plus Ablation (N=9)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 25 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 5 | 1
Blurred vision (Eye disorders) | 0 | 1
Burn (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Chills (General disorders) | 3 | 0
Colitis (General disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 2 | 0
Conjunctivitis (Infections and infestations) | 3 | 0
Constipation (Gastrointestinal disorders) | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Depression (Psychiatric disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 12 | 0
Dizziness (Nervous system disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 1
Dry eye (Eye disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 17 | 8
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 3 | 0
Floaters (Eye disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 4 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Metabolism and nutrition disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Pain (General disorders) | 6 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Prostratic obstruction (Reproductive system and breast disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 5
Restlessness (Nervous system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 2
Watering eyes (Eye disorders) | 0 | 1
Weight loss (Investigations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT02437071/Prot_SAP_000.pdf